CLINICAL TRIAL: NCT02416544
Title: The Effectiveness of Low Calorie Low Salt Lunch for Weight Reduction of Workers of a Health Promoting Hospital
Acronym: HPH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Ju Young Kim, Clinical Assistant Professor, Seoul National University Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: B-1403-244-005; B-1403-244-005 (Other: SeoulNUH)
Record Dates: First submitted 2014-04-20; First posted 2015-04-15 (Estimated); Last update posted 2015-04-15 (Estimated); Status verified 2015-04

CONDITIONS: Overweight; Obesity
Keywords: Overweight; Obesity; Caloric Restriction; Diet, Reducing; Diet, Sodium-Restricted; Body Weight Changes; Energy intake; Feeding Behavior
MeSH Terms: conditions — Overweight; Obesity; Body Weight Changes; Feeding Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Full participation (Experimental): Participants in this group receive lunch which is calorie-restricted and low-salt during 12 weeks, the total duration of this study.
  Interventions: Other: Lunch which is calorie-restricted and low-salt
- Two thirds participation (Experimental): Participants in this group starts lunch which is calorie-restricted and low-salt after 4 weeks from the beginning of the study and maintain the diet during 8 weeks.
  Interventions: Other: Lunch which is calorie-restricted and low-salt
- One thirds participation (Experimental): Participants in this group starts lunch which is calorie-restricted and low-salt after 8 weeks from the beginning of the study and maintain the diet during 4 weeks.
  Interventions: Other: Lunch which is calorie-restricted and low-salt

INTERVENTIONS:
Other: Lunch which is calorie-restricted and low-salt — Comparison of different duration of feeding lunch which is calorie-restricted and low-salt

SUMMARY:
The aim of this study is to evaluate the effectiveness of Low Calorie Low Salt Lunch for Weight Reduction in overweight or obese workers of a health promoting hospital.

ELIGIBILITY:
Inclusion Criteria:

* Overweight or obese
* Hospital workers

Exclusion Criteria:

* History of major medical problems such as heart disease in the last 6 months
* Orthopaedic or joint problems that would be a barrier to physical activity
* Pregnancy
* Recent weight change of ≥10% of baseline weight
* Taking medications that might affect body weight
* Participation in other program about weight control
* Alcohol or substance abuser
* Other uncontrolled psychiatric problems
* Eating disorders

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2014-04; Primary Completion 2014-09 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline in weight | 4 weeks, 8 weeks, and 12 weeks
  Participants will be monitored for up to 12 weeks after intervention

SECONDARY OUTCOMES:
Change from baseline in waist circumference | 4 weeks, 8 weeks, and 12 weeks
  Participants will be monitored for up to 12 weeks after intervention

OTHER OUTCOMES:
Total calorie with sodium intake by 24 hour recall assessment | Baseline, 4 weeks, 8 weeks, and 12 weeks
  Participants will be monitored for up to 12 weeks after intervention
Personal history of weight change | Baseline and 12 weeks
  Questionnaire about personal history of weight change
Smoking (Questionnaire) | Baseline and 12 weeks
  Questionnaire about smoking behavior
Alcohol intake (Questionnaire) | Baseline and 12 weeks
  Questionnaire about the frequency and amount of drinking
Stress status (Questionnaire) | Baseline and 12 weeks
  Questionnaire about stress status
Physical activities (Questionnaire) | Baseline and 12 weeks
  Questionnaire about the frequency and intensity of physical activities
Eating habits (Questionnaire) | Baseline and 12 weeks
  Eating habits will be assessed by asking how often participants eat breakfast and intake different food groups such as fruits, vegetables, dairy products, noodles, cereals, fish, pork, meat products, carbonated beverages and tofu.
Satisfaction regarding low calorie low salt lunch (Questionnaire) | Baseline and 12 weeks
  Questionnaire about satisfaction, acceptance and proposition.

CONTACTS AND LOCATIONS:
Overall Officials: Ju Young Kim, MD. PhD., Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

REFERENCES:
- [Background] Morgan PJ, Collins CE, Plotnikoff RC, Cook AT, Berthon B, Mitchell S, Callister R. Efficacy of a workplace-based weight loss program for overweight male shift workers: the Workplace POWER (Preventing Obesity Without Eating like a Rabbit) randomized controlled trial. Prev Med. 2011 May;52(5):317-25. doi: 10.1016/j.ypmed.2011.01.031. Epub 2011 Feb 20. PMID 21300083
- [Background] Groene O, Jorgensen SJ. Health promotion in hospitals--a strategy to improve quality in health care. Eur J Public Health. 2005 Feb;15(1):6-8. doi: 10.1093/eurpub/cki100. No abstract available. PMID 15788796
- [Background] Handley MA, Schillinger D, Shiboski S. Quasi-experimental designs in practice-based research settings: design and implementation considerations. J Am Board Fam Med. 2011 Sep-Oct;24(5):589-96. doi: 10.3122/jabfm.2011.05.110067. PMID 21900443
- See also: World Health Organization, regional office for europe — http://www.euro.who.int/en/home